CLINICAL TRIAL: NCT06102993
Title: Characterization of New Serum Biomarkers of Ferroptosis in Patients With COPD With/Without Risk of Cardiovascular Events. Pathophysiological Implications, Diagnostics and Prognoses. FerrEPOC Study
Brief Title: Ferroptosis in Patients With COPD COPD With/Without Risk of Cardiovascular Events. Pathophysiological Implications, Diagnostics and Prognoses. FerrEPOC Study.
Acronym: FerrEPOC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Carlos Antonio Amado Diago, MD PhD, Hospital Universitario Marqués de Valdecilla
Other Study IDs: 2023.297
Record Dates: First submitted 2023-10-21; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: COPD Exacerbation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- COPD GOLD 1
  Interventions: Other: Non-interventional study
- COPD GOLD 2
  Interventions: Other: Non-interventional study
- COPD GOLD 3
  Interventions: Other: Non-interventional study
- COPD GOLD 4
  Interventions: Other: Non-interventional study
- Control group
  Interventions: Other: Non-interventional study
- Exacerbated COPD
  Interventions: Other: Non-interventional study

INTERVENTIONS:
Other: Non-interventional study — The only intervention is to analyze serum molecules of patients with COPD and controls without COPD.

SUMMARY:
Iron metabolism is related to several biochemical and functional factors that have a mayor impact in chronic obstructive pulmonary disease (COPD) such as hypoxia, hypercapnia, oxidative stress, chronic inflammation, cellular senescence, sarcopenia and ferroptosis. Ferroptosis is a specific form of cell death induced by excess intracellular free iron that generates lipid peroxidation of cell membranes, with subsequent cell death. The existence of excess ferroptosis in COPD due to tobacco smoke has been widely demonstrated in vitro both in respiratory tissue and in skeletal muscle. Iron and lipid metabolism disorders are an essential part of the pathogenesis of ferroptosis. These disorders have also been related to diseases that occur concomitantly with COPD, such as cardiovascular diseases. Recently, new genes related to iron metabolism that are involved in the development of ferroptosis have been identified. Proteins related with these genes have not been studied in vivo in the context of COPD and cardiovascular diseases. Some of them are purely intracellular in expression, but the expression of some of them can be measured in blood using methods available to any clinical laboratory. After an exhaustive study of the literature, we have selected a small group of circulating proteins expressed in DEGs (Differentially Expressed Genes) related to ferroptosis that overlap with the DEGs of COPD and the DEGs of atherosclerosis to evaluate the relationship between these molecules and clinical variables of COPD and their potential utility in identifying the risk of exacerbations, admissions, and cardiovascular events in COPD. This study could identify a trait in COPD useful for selecting patients at greater risk of exacerbation due to the relationship between ferroptosis and systemic inflammation and oxidative stress, cardiovascular risk and, in general, a worse prognosis of the disease. In addition, the identification of this trait can have important therapeutic implications.

ELIGIBILITY:
Patients with stable phase COPD (not exacerbated) diagnosed according to GesePOC criteria (Spanish guidelines of COPD), over 40 years of age (patients with a history of smoking and forced spirometry after a BD test with a quotient of 0.7) will be included. These patients may or may not have clinical atherosclerosis with/without CCV risk factors and will be studied globally and in groups. The group of acute COPD will consist of patients who have been admitted to the pneumology service diagnosed with exacerbation of COPD syndrome. They must have been diagnosed with COPD according to the GesEPOC (Spanish guidelines of COPD) criteria prior to admission. The control group will consist of 30-40 active smoking volunteers or former smokers without COPD matched by age, level of smoking, without respiratory or renal diseases or serious chronic conditions (severe, known HF, malignant diseases in progression...). COPD will be ruled out by spirometry and the rest of

the pathology will be ruled out by means of a clinical interview and review of ancient history. Stable-phase COPD who have renal failure (Glomerular filtration estimated by the CDK-EPI formula of less than 60 ml/min/1.73 m2), stable phase COPD who have undergone respiratory rehabilitation for at least 6 months before entering the study, or COPD in a stable phase with other diseases or drugs that may cause alterations in the parameters studied (specifically: active tumor diseases, sepsis, critical situations from another origin) will be excluded. Although a group of patients with iron deficiency anemia or iron deficiency without anemia will be included, we do not expect MIFRP to have prognostic utility in this group, so patients with iron deficiency anemia will be excluded from the prospective part of the study, according to the work of Pérez-Peiró et al. (11).

Patients in the COPD group in the stable phase will be followed for one year in outpatient pneumology clinics. During the follow-up, all researchers related to the follow-up will not know the results of the blood samples. During this time, patients with respiratory exacerbation will go to the Emergency Department freely, and a team of doctors not related with the study will decide whether or not to hospitalize patients according to their own clinical criteria.

Ages: 40 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Ambispective Observational Cohort Study to be carried out at the Marqués de Valdecilla University Hospital in Santander (Spain). Patients will be recruited successively among those who attend the outpatient clinic for COPD, smoking cessation in Pulmonology and among those who go to the Emergency Department and are going to be admitted due to an exacerbation of COPD.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Time to hospitalization | 1 year after entering the study

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Marqués de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No